CLINICAL TRIAL: NCT03125343
Title: A Multicenter Prospective National Cohort Study for Patients With Advanced Rectal Cancer - is it Possible to Induce Remission and Avoid Surgery - Watch and Wait?
Brief Title: Watch and Wait as Treatment for Patients With Rectal Cancer
Acronym: WoW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Angenete, M.D, Ph.D., Sahlgrenska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WoW
Record Dates: First submitted 2017-03-20; First posted 2017-04-24 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Rectal Neoplasms
Keywords: radiotherapy; chemotherapy; complete response
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Endoscopy; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: All patients with complete response defined as described above will be offered to enter the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No surgery (Experimental): Patients with indication of complete response on follow-up MRI will undergo endoscopy, and digital rectal examination to ascertain complete response. MRI together with documentation from endoscopy will be reviewed at the Regional University Hospital to establish agreement regarding interpretation.
  Interventions: Procedure: endoscopy; Device: MRI
- Surgery (Active Comparator): Patients with indication of complete response on follow-up MRI will undergo endoscopy, and digital rectal examination to ascertain complete response. MRI together with documentation from endoscopy will be reviewed at the Regional University Hospital to establish agreement regarding interpretation. Patients with complete response will be offered watch and wait strategy, but the patients that want surgery will be operated according to the multi disciplinary conference decision.
  Interventions: Procedure: Surgery; Device: MRI

INTERVENTIONS:
Procedure: endoscopy — Continuous follow-up. All patients with complete response will be followed for ten years. Details from the follow-up schedule will be registered in clinical record forms including information on the endoscopic findings, MRI findings and digital examination.
  They will be followed ever third month for the first two years as follows:
  * PET-CT is optional, but can be performed at inclusion
  * Pelvic MRI including diffusion weighted imaging according to appendix C.
  * Clinical examination
  * Endoscopy (flexible sigmoidoskopy) with photodocumentation
  * CEA
  After two years the patients will be followed every six month with:
  * Pelvic MRI including diffusion weighted imaging according to appendix as at baseline
  * Clinical examination
  * Endoscopy with photodocumentation
  * CEA
  Arms: No surgery
Procedure: Surgery — Surgery according to recommendations from the multidisciplinary group in patients that prefer surgery to a watch and wait strategy
  Arms: Surgery
Device: MRI

SUMMARY:
A national cohort study with all patients scheduled for neoadjuvant treatment with (chemo)radiotherapy or short course radiotherapy with delayed surgery 6-8 weeks) for rectal cancer staged as cT4bNX/anycTanycN and cMRF+/anycTanycN and lateral lymph nodes on MRI (and patients that have been offered short course raditotherapy with delayed surgery due to various reasons). The tumours are positioned midrectal or low and are palpable with the finger. The patients offered this treatment after recommendations on their local multidisciplinary tumour board will be will be informed and offered to participate in the study. Patients scheduled for short course radiotherapy with immediate surgery cannot be included.

DETAILED DESCRIPTION:
• Biopsies and blood from patients with rectal cancer subject to neoadjuvant treatment with (chemo)radiotherapy or radiotherapy 5x5 Gy with at least 6-8 weeks wait until surgery. All patients will be asked to answer a QoL questionnaire (appendix C) to cover their experiences of the neaodajvuant treatment. (Answered at diagnosis and at evaluation of treatment and decision of surgery or inclusion in the Watch and Wait part of the study).

All patients will undergo scheduled (chemo)radiotherapy according to national guidelines. The patients with chemoradiotherapy will be evaluated at 8-10 weeks after completed treatment (25) with pelvic MRI. After this evaluation at 8-10 weeks patients with suspected complete response or near complete response will examined according to the protocol below.

All patients that are considered to have complete response will be offered a "Watch and wait" approach with follow-up according to the protocol. They will then be followed at one of the Regional University Hospitals within their catchment are.

All patients with a palpable rectal cancer staged as cT4bNX/anycTanycN and cMRF+/anycTanycN and lateral lymph nodes on MRI (and patients that have been offered short course raditotherapy with delayed surgery due to various reasons) that does not achieve complete response will serve as control and will be treated with surgery as planned prior to initiation of (chemo)radiotherapy.

Patients with indication of complete response on follow-up MRI will undergo endoscopy, and digital rectal examination to ascertain complete response. MRI together with documentation from endoscopy will be reviewed at the Regional University Hospital to extablish agreement regarding interpretation. All the below mentioned criteria must be fullfilled to be considered complete response:

1. No suspicious metastatic lymph nodes or evidence of remaining tumour on MRI. In the majority of cases a complete response on MRI will be seen as areas of homogeneous fibrosis. Absence of any remaining pathological tissue is seen in a minority of cases.
2. Endoscopic examination with light/white mucosa or scar, telangiectasies. Prescence of fibrosis and oedema.
3. No palpable tumour on clinical examination (26).

In the spring of 2023 200 pts included. An amendment was sent to the ethical review board to enable continued inclusion while the initial 200 pts are analyzed. This has been approved and the study has thus planned continuation for another 2-3 years.

ELIGIBILITY:
Inclusion Criteria:

All patients in Sweden with a palpable rectal cancer staged as cT4bNX/anycTanycN and cMRF+/anycTanycN and lateral lymph nodes on MRI considered appropriate for 5x5 Gy and 6-8 weeks of wait prior to surgery according to Stockholm III (28) or a palpable rectal cancer staged as cT4bNX/anycTanycN and cMRF+/anycTanycN and lateral lymph nodes on MRI a planned schedule for CRT according to the Swedish National Program for rectal cancer scheduled for neoadjuvant therapy are possible to include.

The study includes two parts, where part one is optional in including hospitals. The aim of the biopsy substudy to identify tumour and plasma markers for complete response, thus all patients that will receive (chemo)radiotherapy in the neoadjuvant setting are included to provide a control for the biopsies.

For the WoW part of the study all patients that achieve complete response after neoadjuvant treatment according to the specified criteria above can be included in the Watch and Wait protocol. In detail this includes patients with:

Midrectal or low rectal cancers that are palpable and considered with an indication of 5x5 Gy and long wait (6-8 weeks) (the indication for waiting may be logistics, co-morbidity, advanced age):

* cT4bNX
* anycTanycN and cMRF+ anycTanycN and lateral lymph nodes on MRI

Exclusion Criteria:

* No informed consent received for participation.
* Patients with rectal cancer that is scheduled for (chemo) radiotherapy but is not palpable during rectal examination (10-15 cm) as this cannot be examined by digital examination and followed as scheduled.
* Contraindication for MRI such as presence of non compatible metallic implants or claustrophobia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival. | 3 years
  Thus this includes patients that have had regrowth and been operated for their tumour. Includes metastastic surgery as well

SECONDARY OUTCOMES:
Percentage re-growth during follow-up | 10 years
  Endoscopic or MRI indication of regrowth
Local recurrence after salvage surgery due to regrowth | 10 years
  Local recurrence as shown by MRI, endoscopy or digital examination
Results after surgery for re-growth | 10 years
  Complications and mortality after surgery
Long-term survival | 10 years
  Overall survival
Number of patients with no response, partial response and complete response. | Accrual period - probably 4 years
  Number of patients in each group - no response, partial response and complete response
Anorectal function measured by LARS score | 5 years
  Anorectal function measured by LARS and then compared to patients operated.
Quality of life measured by a clinometric approach | up to 24 months
  QoL measurments sent to patients
Health economic evaluation | 5 years
  A cost efficiency analysis

CONTACTS AND LOCATIONS:
Overall Officials: Eva Angenete, M.D., Ph.D., Principal Investigator — Sahlgrenska Academy at Gothenburg University
Locations (2):
- Sweden (2):
  - Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg
  - Karolinska Institutet, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided